CLINICAL TRIAL: NCT02904096
Title: Radiesse® Post Approval Safety Study For the Treatment of Hands With Moderate to Very Severe Dorsal Volume Loss
Brief Title: Radiesse® Safety Study For the Treatment of Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P151009, M900311002
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-01

CONDITIONS: Volume Loss in the Dorsum of the Hand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- "Grade 4 Hands" group (Experimental): "Grade 4 Hands" group will be subjects with hand grading of grade 4 (very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand). "Grade 4 Hands" group subjects will receive Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment. Subjects in "Grade 4 Hands" group can have up to three retreatments over an 18 month period.
  Interventions: Device: Radiesse injectable implant and 2% lidocaine HCL
- "Grade 2 or 3 Hands" group (Experimental): "Grade 2 or 3 Hands" group will be subjects with hand grading of grade 2 or grade 3 (moderate to severe loss of fatty tissue, mild to moderate visibility of veins and tendons in the dorsal hand). "Grade 2 or 3 Hands" group subjects will receive Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment. Subjects in "Grade 2 or 3 Hands" group can have up to three retreatments over an 18 month period.
  Interventions: Device: Radiesse injectable implant and 2% lidocaine HCL

INTERVENTIONS:
Device: Radiesse injectable implant and 2% lidocaine HCL — Radiesse injectable implant injected in small boluses (0.2-0.5cc/bolus). No more than 0.5cc per bolus. No more than 3 cc (2 syringes) will be injected per hand.

SUMMARY:
The primary objective of this study is to evaluate the safety of Radiesse implantation for very severe volume loss in the dorsum of the hand at 6 months after treatment.

DETAILED DESCRIPTION:
This is a 2-year post approval safety (PAS) study evaluating the Adverse Event (AE) rate of Merz Hand Grading Scale (MHGS) baseline grade 4 hands (Group A) compared to the AE rate of MHGS baseline grade 2-3 hands (Group B).

Subjects will be recruited at each site with the intention to have an equal number of subjects in Group A and Group B. All subjects will receive an initial Radiesse hand treatment in both hands, and up to 3 retreatments in the study. Hands will be assessed by evaluators on the MHGS who will be blinded to group, treatment details, time since last treatment, and number of retreatments.

ELIGIBILITY:
Inclusion Criteria:

1. Has hands rating 2, 3, or 4 on the validated MHGS as determined by a live, masked evaluator.
2. Is at least 22 years of age.
3. Understands and accepts the obligation not to receive any other procedures in the dorsum of the hands through the end of the study.
4. Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits and meet all study requirements.

Exclusion Criteria:

1. Was a participant in the Radiesse hands pre-market clinical study
2. Has been treated with fat injections or Radiesse in the hands, has hand deformities, or has received surgery in the dorsum of the hands.
3. Has any medical condition with the potential to interfere with the study or increase the risk of AEs.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (9):
- United States (9):
  - Merz Investigative Site #0010393, Sacramento, California
  - Merz Investigative Site #0010321, San Diego, California
  - Merz Investigative Site #0010358, Vista, California
  - Merz Investigative Site #0010099, West Hollywood, California
  - Merz Investigative Site #0010405, New York, New York
  - Merz Investigative Site #0010406, New York, New York
  - Merz Investigative Site #0010322, Austin, Texas
  - Merz Investigative Site #0010125, Plano, Texas
  - Merz Investigative Site #0010392, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 investigational sites in the United States.
Pre-assignment Details: A total of 256 subjects were enrolled and treated, out of which 216 subjects completed the study.
Groups:
- Group A: MHGS Grade 4 Hands Group: Subjects with Merz hand grading scale (MHGS) Grade 4, which indicates very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2 percent (%) lidocaine hydrochloric acid (HCL) up to 3 cubic centimeter (cc) (2 syringes) per hand per treatment at Day 0 (Screening or Enrollment). All subjects were treated in the dorsum of the hands. Based on the investigator and subject's decision, subjects received up to three retreatments at Months 6, 12, and 18.
- Group B: MHGS Grade 2 or 3 Hands Group: Subjects with MHGS Grade 2 or 3, which indicates moderate to severe loss of fatty tissue and mild to moderate visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment at Day 0 (Screening or Enrollment). All subjects were treated in the dorsum of the hands. Based on the investigator and subject's decision, subjects received up to three retreatments at Month 6, 12, and 18.
Period: Overall Study
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Started | 130 | 126
Completed | 111 | 105
Not Completed | 19 | 21
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 10 | 17
Not completed — Non-compliant | 3 | 1
Not completed — Sponsor instructed | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all subjects who were exposed to the study device at enrollment.
Groups:
- Group A: MHGS Grade 4 Hands Group: Subjects with MHGS Grade 4, which indicates very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment at Day 0 (Screening or Enrollment). All subjects were treated in the dorsum of the hands. Based on the investigator and subject's decision, subjects received up to three retreatments at Months 6, 12, and 18.
- Total: Total of all reporting groups
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group | Total
Number analyzed (Participants) | 130 | 126 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 107 | 178
  >=65 years | 59 | 19 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 118 | 246
  Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 123 | 118 | 241
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 122 | 117 | 239
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 126 | 256
Fitzpatrick skin type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Type I | 13 | 12 | 25
    Type II | 63 | 65 | 128
    Type III | 38 | 39 | 77
    Type IV | 11 | 7 | 18
    Type V | 3 | 0 | 3
    Type VI | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Device-and/or Injection-related Severe Treatment-emergent Adverse Events (TEAEs) in the Grade 4 Hands Group Versus the Grade 2-3 Hands Group at Month 6
Description: Proportion refers to percentage of subjects with device-and/or injection-related severe TEAEs.
Time Frame: Month 6
Population: The SES was the subset of all subjects who were exposed to the study device at enrollment.
Measure: Number; unit: percentage of subjects
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 130 | 126
percentage of subjects | 1.5 | 0
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group vs Group B: MHGS Grade 2 or 3 Hands Group; Test type: Non-Inferiority — Estimates for PA, PB, and PA-PB were reported together with one-sided 95% confidence interval (CI) for PA-PB constructed via the Farrington-Manning likelihood method. Here PA and PB are the percentage of subjects in Group A and B (Non-inferiority margin = 12%); Difference in percentage = 1.5, 95% CI 1-sided [upper limit 3.35]

2. Secondary Outcome: Proportion of Subjects With Device-and/Injection-related Severe TEAEs in the Grade 4 Hands Group Versus the Grade 2-3 Hands Group at Month 24
Description: Proportion refers to percentage of subjects with device-and/injection-related severe TEAEs.
Time Frame: Month 24
Population: The SES was the subset of all subjects who were exposed to the study device at enrollment.
Measure: Number; unit: percentage of subjects
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 130 | 126
percentage of subjects | 1.5 | 0
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group vs Group B: MHGS Grade 2 or 3 Hands Group; Test type: Other; Difference in Percentage = 1.5, 95% CI 1-sided [upper limit 3.35]

3. Secondary Outcome: Change From Baseline in Range of Motion (ROM) Flexion and Extension (Angle) for Metacarpophalangeal Joints in Each Hand at Month 24
Description: The ROM was assessed using a Jamar finger goniometer. This test passively and actively measured the angle of motion of all five metacarpophalangeal joints in each hand right and left by determining the flexion and extension angles. The flexion determined how far each finger could be flexed at the metacarpophalangeal joint toward the palm. The extension determined how each finger could be extended at the metacarpophalangeal joint away from the palm. Degree scale ranges from 0 to 180 degree. Lower values in flexion angle and extension angle means more deterioration in hand function.
Time Frame: Baseline, Month 24
Population: The SES was the subset of all subjects who were exposed to the study device at enrollment. The SES were evaluable for this measure at a given time period and were included in the assessment.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 112 | 105
degrees
  Change at Month 24, Flexion: Left Hand | 4.10 (10.72) | 2.07 (10.88)
  Change at Month 24, Flexion: Right Hand | 4.20 (10.50) | 3.17 (9.16)
  Change at Month 24, Extension: Left Hand | 1.83 (9.74) | -0.32 (11.88)
  Change at Month 24, Extension: Right Hand | 2.88 (9.98) | 0.72 (13.01)
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Flexion (Left Hand)-baseline and Group A: Flexion (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 2: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Flexion (Right Hand)-baseline and Group A: Flexion (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 3: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Flexion (Left Hand)-baseline and Group B: Flexion (Left Hand)-change from baseline at Month 24; Test type: Other; p = .054, t-test, 1 sided
Statistical Analysis 4: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Flexion (Right Hand)-baseline and Group B: Flexion (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 5: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Extension (Left Hand)-baseline and Group A: Extension (Left Hand)-change from baseline at Month 24; Test type: Other; p = .049, t-test, 1 sided
Statistical Analysis 6: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Extension (Right Hand)-baseline and Group A: Extension (Right Hand)-change from baseline at Month 24; Test type: Other; p = .003, t-test, 1 sided
Statistical Analysis 7: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Extension (Left Hand)-baseline and Group B: Extension (Left Hand)-change from baseline at Month 24; Test type: Other; p = .781, t-test, 1 sided
Statistical Analysis 8: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Extension (Right Hand)-baseline and Group B: Extension (Right Hand)-change from baseline at Month 24; Test type: Other; p = .573, t-test, 1 sided

4. Secondary Outcome: Change From Baseline in Functional Dexterity in Each Hand at Month 24
Description: The functional dexterity test (FDT) assessed the fine motor skills (dexterity) that means it assessed the subject's ability to use the hand for daily tasks requiring the 3-jaw chunk prehensions that is buttoning, tying shoelaces, screwing a nut and bolt, and lacing yarn using a 16-hole peg board. Functional Dexterity was measured by noting the time in seconds on stopwatch for a hand to invert pegs on a 16-hole pegboard and this test assessed the ability to use hand for daily tasks. Longer times to complete the functional dexterity test means deterioration in hand function.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 112 | 105
seconds
  Change at Month 24: Left Hand | -6.29 (13.50) | -3.76 (4.82)
  Change at Month 24: Right Hand | -4.53 (7.90) | -3.89 (5.34)
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: (Left Hand)-baseline and Group A: (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 2: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: (Right Hand)-baseline and Group A: (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 3: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: (Left Hand)-baseline and Group B: (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 4: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: (Right Hand)-baseline and Group B: (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided

5. Secondary Outcome: Change From Baseline in Sensation to Filament Size Between Metacarpals in Each Hand at Month 24
Description: Sensation in the dorsum of each hand was conducted using a Semmes-Weinstein monofilament touch test. This was assessed using an index finger touch protocol, where by study subject was asked to report when a 2 to 3 centimeter (cm) light touch is felt at 3 different areas of the dorsum of each hand. Sensation results were coded for analysis such as response to 2.83 filament = 1, response to 3.61 filament = 2, response to 4.31 filament = 3, response to 4.56 filament = 4, response to 6.65 filament = 5, and no response to either filament = 6. For sensation testing a value of 1 (response to 2.83 filament) is considered normal while a value of 2 (response to 3.61) would show diminished light touch. Score ranges from 1 to 6. A higher value in sensation measurements is associated with a deterioration in hand function.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 112 | 105
scores on a scale
  Change at Month 24: Left Hand | -0.52 (0.60) | -0.44 (0.60)
  Change at Month 24: Right Hand | -0.49 (0.64) | -0.52 (0.64)
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: (Left Hand)-baseline and Group A: (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 2: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: (Right Hand)-baseline and Group A: (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 3: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: (Left Hand)-baseline and Group B: (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 4: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: (Right Hand)-baseline and Group B: (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided

6. Secondary Outcome: Change From Baseline in Grip Strength, Tip Pinch Strength, Key Pinch Strength, and Palmar Strength in Each Hand at Month 24
Description: Hand strength was assessed in two ways grip and pinch strengths. Grip strength was assessed using a standard, adjustable-handle Jamar hydraulic hand dynamometer. Pinch strength was assessed in three different ways such as tip (two-point) pinch, key (lateral) pinch, and palmar (three-jaw chuck) pinch using the Jamar hydraulic pinch gauge. Lower values (pounds) in hand grip and pinch strength are associated with deterioration in function.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 112 | 105
pounds
  Change at Month 24, Grip Strength: Left Hand | -3.63 (8.68) | -4.65 (11.17)
  Change at Month 24, Grip Strength: Right Hand | -2.28 (7.36) | -3.37 (10.85)
  Change at Month 24, Tip Pinch Strength: Left Hand | 1.26 (2.94) | 1.70 (3.21)
  Change at Month 24, Tip Pinch Strength: Right Hand | 1.60 (2.99) | 1.46 (3.48)
  Change at Month 24, Key Pinch Strength: Left Hand | 0.90 (2.88) | 1.12 (2.76)
  Change at Month 24, Key Pinch Strength: Right Hand | 1.33 (2.99) | 1.26 (2.99)
  Change at Month 24,Palmar Pinch Strength:Left Hand | 0.68 (2.78) | 0.43 (3.21)
  Change at Month 24,PalmarPinch Strength:Right Hand | 0.54 (3.04) | 0.40 (3.04)
Statistical Analysis 1: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand grip strength (Left Hand)-baseline and Group A: Hand grip strength (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 2: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand grip strength (Right Hand)-baseline and Group A: Hand grip strength (Right Hand)-change from baseline at Month 24; Test type: Other; p = .001, t-test, 1 sided
Statistical Analysis 3: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand grip strength (Left Hand)-baseline and Group B: Hand grip strength (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 4: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand grip strength (Right Hand)-baseline and Group B: Hand grip strength (Right Hand)-change from baseline at Month 24; Test type: Other; p = .002, t-test, 1 sided
Statistical Analysis 5: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand tip pinch strength (Left Hand)-baseline and Group A: Hand tip pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 6: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand tip pinch strength (Right Hand)-baseline and Group A: Hand tip pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 7: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand tip pinch strength (Left Hand)-baseline and Group B: Hand tip pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 8: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand tip pinch strength (Right Hand)-baseline and Group B: Hand tip pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 9: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand key pinch strength (Left Hand)-baseline and Group A: Hand key pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p = .001, t-test, 1 sided
Statistical Analysis 10: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand key pinch strength (Right Hand)-baseline and Group A: Hand key pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 11: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand key pinch strength (Left Hand)-baseline and Group B: Hand key pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 12: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand key pinch strength (Right Hand)-baseline and Group B: Hand key pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p < .001, t-test, 1 sided
Statistical Analysis 13: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand palmar pinch strength (Left Hand)-baseline and Group A: Hand palmar pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p = .010, t-test, 1 sided
Statistical Analysis 14: Comparison: Group A: MHGS Grade 4 Hands Group; Comparison between Group A: Hand palmar pinch strength (Right Hand)-baseline and Group A: Hand palmar pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p = .060, t-test, 1 sided
Statistical Analysis 15: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand palmar pinch strength (Left Hand)-baseline and Group B: Hand palmar pinch strength (Left Hand)-change from baseline at Month 24; Test type: Other; p = .177, t-test, 1 sided
Statistical Analysis 16: Comparison: Group B: MHGS Grade 2 or 3 Hands Group; Comparison between Group B: Hand palmar pinch strength (Right Hand)-baseline and Group B: Hand palmar pinch strength (Right Hand)-change from baseline at Month 24; Test type: Other; p = .177, t-test, 1 sided

7. Secondary Outcome: Number of Subjects With MHGS Scores Greater Than or Equal (>=) to 1-point Improvement From Baseline in Both Hands at Month 3 After Initial Treatment
Description: The MHGS was used to measure clinical effectiveness of the Radiesse hand treatments by a masked evaluator performing live, dorsal hand assessments. The MHGS was an ordinal scale; therefore, ratings were made at a single, live rating at a specific study time point. A measure of successful or improved treatment effect was demonstrated by a decrease in MHGS score. MHGS had 5 categories, where: 0 (no loss of fatty tissue); 1 (mild loss of fatty tissue; slight visibility of veins); 2 (moderate loss of fatty tissue; mild visibility of veins and tendons); 3 (severe loss of fatty tissue; moderate visibility of veins and tendons); 4(very severe loss of fatty tissue; marked visibility of veins and tendons).
Time Frame: Month 3
Population: The SES was the subset of all subjects who were exposed to the study device at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 130 | 126
Participants | 117 | 104

8. Secondary Outcome: Number of Subjects With MHGS >=1-point Improvement Following 3 Months After Retreatment at Months 9, 15 and 21
Description: as for outcome 7
Time Frame: Months 9, 15, and 21
Population: Data were not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Subjects With Any Improvement on Global Aesthetic Improvement Scale (GAIS) From Baseline in Both Hands at Month 3 After Initial Treatment
Description: The GAIS is a 7-point scale. The 7-point scale are as follow: +3 (very much improved), +2 (much improve), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), and -3 (very much worse).
Time Frame: Month 3
Population: The SES was the subset of all subjects who were exposed to the study device at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 130 | 126
Participants | 115 | 118

10. Secondary Outcome: Number of Subjects With Any Improvement on GAIS Following 3 Months After Retreatment at Months 9, 15 and 21
Description: as for outcome 9
Time Frame: Months 9, 15, and 21
Population: Data were not collected and analyzed for this outcome measure due to change in planned analysis.
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: The investigator asked the subject for adverse events (AEs) systematically at each visit.
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
All-Cause Mortality (participants affected / at risk) | 1/130 | 0/126
Serious Adverse Events (participants affected / at risk) | 9/130 | 3/126
Other Adverse Events (participants affected / at risk) | 70/130 | 57/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: MHGS Grade 4 Hands Group (N=130) | Group B: MHGS Grade 2 or 3 Hands Group (N=126)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 1
Sarcoma excision (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: MHGS Grade 4 Hands Group (N=130) | Group B: MHGS Grade 2 or 3 Hands Group (N=126)
Injection site bruising (General disorders) | 39 | 37
Nodule (General disorders) | 17 | 14
Pain (General disorders) | 11 | 9
Swelling (General disorders) | 32 | 27
Erythema (Skin and subcutaneous tissue disorders) | 20 | 8
Haematoma (Vascular disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02904096/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT02904096/SAP_001.pdf